CLINICAL TRIAL: NCT00585195
Title: PHASE 1 SAFETY, PHARMACOKINETIC AND PHARMACODYNAMIC STUDY OF PF-02341066, A MET/HGFR SELECTIVE TYROSINE KINASE INHIBITOR, ADMINISTERED ORALLY TO PATIENTS WITH ADVANCED CANCER
Brief Title: A Study Of Oral PF-02341066, A C-Met/Hepatocyte Growth Factor Tyrosine Kinase Inhibitor, In Patients With Advanced Cancer
Acronym: PROFILE 1001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081001; PROFILE 1001 (Other: Alias Study Number)
Record Dates: First submitted 2007-12-29; First posted 2008-01-03 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Non-Small Cell Lung Cancer ALK-positive; Non-Small Cell Lung Cancer c-Met Dependent; Non-Small Cell Lung Cancer ROS Marker Positive; Systemic Anaplastic Large-Cell Lymphoma; Advanced Malignancies Except Leukemia
Keywords: Crizotinib; dose-finding; drug-drug interaction; ALK rearrangements; c-Met mutations or amplifications; c-Met dependent tumors; ROS1 rearrangements; c-Met exon 14 deletion; c-Met exon 14 skipping; c-Met exon 14 alterations
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Crizotinib; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-02341066; Drug: Rifampin; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-02341066 — Escalating doses of PF-02341066 will be administered orally on a continuous dosing schedule. Doses to be evaluated will range from 50 mg to 2000 mg/day administered either once or twice a day. A treatment cycle is considered to be 28 days (or 21 days depending on the cohort).
Drug: Rifampin — 600 mg QD administered from Cycle 1, Day 16 to Cycle 2, Day 1 (14 days of dosing) in combination with PF-02341066.
Drug: Itraconazole — Multiple Dose Design: 200 mg QD administered from Cycle 1, Day 1 to Cycle 1, Day 16 (16 days) in combination with PF-02341066.

SUMMARY:
PF-02341066 may work in cancer by blocking the cell growth, migration and invasion of tumor cells. PF-02341066 is a new class of drugs called c-Met/Hepatocyte growth factor receptor tyrosine kinase inhibitors. This compound is also an inhibitor of the anaplastic lymphoma kinase (called ALK) tyrosine kinase and ROS receptor tyrosine kinases. This research study is the first time PF-02341066 will be given to people. PF-02341066 is taken by mouth daily.

ELIGIBILITY:
Inclusion Criteria:

* Advanced malignancies (except leukemias), histologically proven at diagnosis; Histologically confirmed advanced malignancies that are known to be sensitive to PF-03241066 inhibition, e.g. ALK, c-MET and ROS
* Solid tumors must have measurable disease (Recommended Phase 2 Dose Cohort patients with non-measurable disease may enter on a case-by-case basis); not required for DDI sub-studies.
* Adequate blood cell counts, kidney function, liver function and Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 (for the Recommended Phase 2 Cohort, a ECOG score of 2 may be allowed on a case-by-case basis)

Exclusion Criteria:

* Major surgery, radiation therapy or anti-cancer therapy within 2 to 4 weeks of starting study treatment, depending on the patient cohort
* Prior stem cell transplant except of patients with neuroblastoma, lymphoma or myeloma
* Active or unstable cardiac disease or heart attack within 3 months of starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2006-04-19 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (23):
  - University of California, Irvine Medical Center, Orange, California
  - University of Colorado Hospital/ Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Joslin Beetham Eye Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center: Breast and Imaging Center, New York, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Ohio State Eye and Ear Institute, Columbus, Ohio
  - The Ohio State University Martha Morehouse Medical Plaza, Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - The University of Vermont Medical Center, Burlington, Vermont
  - The University of Vermont Cancer Center, Burlington, Vermont
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Japan (3):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kindai University Hospital, Sayama, Osaka
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ng TL, Tsui DCC, Wang S, Usari T, Patil T, Wilner K, Camidge DR. Association of anticoagulant use with clinical outcomes from crizotinib in ALK- and ROS1-rearranged advanced non-small cell lung cancers: A retrospective analysis of PROFILE 1001. Cancer Med. 2022 Dec;11(23):4422-4429. doi: 10.1002/cam4.4789. Epub 2022 May 5. PMID 35510711
- [Derived] Camidge DR, Otterson GA, Clark JW, Ignatius Ou SH, Weiss J, Ades S, Shapiro GI, Socinski MA, Murphy DA, Conte U, Tang Y, Wang SC, Wilner KD, Villaruz LC. Crizotinib in Patients With MET-Amplified NSCLC. J Thorac Oncol. 2021 Jun;16(6):1017-1029. doi: 10.1016/j.jtho.2021.02.010. Epub 2021 Mar 4. PMID 33676017
- [Derived] Solomon BJ, Kim EE, Winter M, Monti K, Tang Y, Wilner KD, Wang S, Ou SI. Ophthalmological assessment of crizotinib in advanced non-small-cell lung cancer. Lung Cancer. 2020 Jul;145:167-172. doi: 10.1016/j.lungcan.2020.04.010. Epub 2020 Apr 28. PMID 32460197
- [Derived] Clark JW, Camidge DR, Kwak EL, Maki RG, Shapiro GI, Chen I, Tan W, Randolph S, Christensen JG, Ozeck M, Tang Y, Wilner KD, Salgia R. Dose-escalation trial of the ALK, MET & ROS1 inhibitor, crizotinib, in patients with advanced cancer. Future Oncol. 2020 Jan;16(1):4289-4301. doi: 10.2217/fon-2019-0653. Epub 2019 Nov 28. PMID 31778074
- [Derived] Shaw AT, Riely GJ, Bang YJ, Kim DW, Camidge DR, Solomon BJ, Varella-Garcia M, Iafrate AJ, Shapiro GI, Usari T, Wang SC, Wilner KD, Clark JW, Ou SI. Crizotinib in ROS1-rearranged advanced non-small-cell lung cancer (NSCLC): updated results, including overall survival, from PROFILE 1001. Ann Oncol. 2019 Jul 1;30(7):1121-1126. doi: 10.1093/annonc/mdz131. PMID 30980071
- [Derived] Camidge DR, Kim EE, Usari T, Polli A, Lewis I, Wilner KD. Renal Effects of Crizotinib in Patients With ALK-Positive Advanced NSCLC. J Thorac Oncol. 2019 Jun;14(6):1077-1085. doi: 10.1016/j.jtho.2019.02.015. Epub 2019 Feb 26. PMID 30822515
- [Derived] Yoneda KY, Scranton JR, Cadogan MA, Tassell V, Nadanaciva S, Wilner KD, Stollenwerk NS. Interstitial Lung Disease Associated With Crizotinib in Patients With Advanced Non-Small Cell Lung Cancer: Independent Review of Four PROFILE Trials. Clin Lung Cancer. 2017 Sep;18(5):472-479. doi: 10.1016/j.cllc.2017.03.004. Epub 2017 Mar 14. PMID 28373069
- [Derived] Shaw AT, Ou SH, Bang YJ, Camidge DR, Solomon BJ, Salgia R, Riely GJ, Varella-Garcia M, Shapiro GI, Costa DB, Doebele RC, Le LP, Zheng Z, Tan W, Stephenson P, Shreeve SM, Tye LM, Christensen JG, Wilner KD, Clark JW, Iafrate AJ. Crizotinib in ROS1-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Nov 20;371(21):1963-71. doi: 10.1056/NEJMoa1406766. Epub 2014 Sep 27. PMID 25264305
- [Derived] Go H, Kim DW, Kim D, Keam B, Kim TM, Lee SH, Heo DS, Bang YJ, Chung DH. Clinicopathologic analysis of ROS1-rearranged non-small-cell lung cancer and proposal of a diagnostic algorithm. J Thorac Oncol. 2013 Nov;8(11):1445-50. doi: 10.1097/JTO.0b013e3182a4dd6e. PMID 24128715
- [Derived] Awad MM, Katayama R, McTigue M, Liu W, Deng YL, Brooun A, Friboulet L, Huang D, Falk MD, Timofeevski S, Wilner KD, Lockerman EL, Khan TM, Mahmood S, Gainor JF, Digumarthy SR, Stone JR, Mino-Kenudson M, Christensen JG, Iafrate AJ, Engelman JA, Shaw AT. Acquired resistance to crizotinib from a mutation in CD74-ROS1. N Engl J Med. 2013 Jun 20;368(25):2395-401. doi: 10.1056/NEJMoa1215530. Epub 2013 Jun 1. PMID 23724914
- [Derived] Camidge DR, Bang YJ, Kwak EL, Iafrate AJ, Varella-Garcia M, Fox SB, Riely GJ, Solomon B, Ou SH, Kim DW, Salgia R, Fidias P, Engelman JA, Gandhi L, Janne PA, Costa DB, Shapiro GI, Lorusso P, Ruffner K, Stephenson P, Tang Y, Wilner K, Clark JW, Shaw AT. Activity and safety of crizotinib in patients with ALK-positive non-small-cell lung cancer: updated results from a phase 1 study. Lancet Oncol. 2012 Oct;13(10):1011-9. doi: 10.1016/S1470-2045(12)70344-3. Epub 2012 Sep 4. PMID 22954507
- [Derived] Ou SH, Azada M, Dy J, Stiber JA. Asymptomatic profound sinus bradycardia (heart rate </=45) in non-small cell lung cancer patients treated with crizotinib. J Thorac Oncol. 2011 Dec;6(12):2135-7. doi: 10.1097/JTO.0b013e3182307e06. PMID 22088989
- [Derived] Shaw AT, Yeap BY, Solomon BJ, Riely GJ, Gainor J, Engelman JA, Shapiro GI, Costa DB, Ou SH, Butaney M, Salgia R, Maki RG, Varella-Garcia M, Doebele RC, Bang YJ, Kulig K, Selaru P, Tang Y, Wilner KD, Kwak EL, Clark JW, Iafrate AJ, Camidge DR. Effect of crizotinib on overall survival in patients with advanced non-small-cell lung cancer harbouring ALK gene rearrangement: a retrospective analysis. Lancet Oncol. 2011 Oct;12(11):1004-12. doi: 10.1016/S1470-2045(11)70232-7. Epub 2011 Sep 18. PMID 21933749
- [Derived] Kijima T, Takeuchi K, Tetsumoto S, Shimada K, Takahashi R, Hirata H, Nagatomo I, Hoshino S, Takeda Y, Kida H, Goya S, Tachibana I, Kawase I. Favorable response to crizotinib in three patients with echinoderm microtubule-associated protein-like 4-anaplastic lymphoma kinase fusion-type oncogene-positive non-small cell lung cancer. Cancer Sci. 2011 Aug;102(8):1602-4. doi: 10.1111/j.1349-7006.2011.01970.x. PMID 21767331
- [Derived] Ou SH, Kwak EL, Siwak-Tapp C, Dy J, Bergethon K, Clark JW, Camidge DR, Solomon BJ, Maki RG, Bang YJ, Kim DW, Christensen J, Tan W, Wilner KD, Salgia R, Iafrate AJ. Activity of crizotinib (PF02341066), a dual mesenchymal-epithelial transition (MET) and anaplastic lymphoma kinase (ALK) inhibitor, in a non-small cell lung cancer patient with de novo MET amplification. J Thorac Oncol. 2011 May;6(5):942-6. doi: 10.1097/JTO.0b013e31821528d3. PMID 21623265
- [Derived] Costa DB, Kobayashi S, Pandya SS, Yeo WL, Shen Z, Tan W, Wilner KD. CSF concentration of the anaplastic lymphoma kinase inhibitor crizotinib. J Clin Oncol. 2011 May 20;29(15):e443-5. doi: 10.1200/JCO.2010.34.1313. Epub 2011 Mar 21. No abstract available. PMID 21422405
- [Derived] Butrynski JE, D'Adamo DR, Hornick JL, Dal Cin P, Antonescu CR, Jhanwar SC, Ladanyi M, Capelletti M, Rodig SJ, Ramaiya N, Kwak EL, Clark JW, Wilner KD, Christensen JG, Janne PA, Maki RG, Demetri GD, Shapiro GI. Crizotinib in ALK-rearranged inflammatory myofibroblastic tumor. N Engl J Med. 2010 Oct 28;363(18):1727-33. doi: 10.1056/NEJMoa1007056. PMID 20979472
- [Derived] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081001&StudyName=A%20Study%20Of%20Oral%20PF-02341066%2C%20A%20c-Met/Hepatocyte%20Growth%20Factor%20Tyrosine%20Kinase%20Inhibitor%2C%20In%20Patients%20With%20Advanced%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a lead-in period of 7 days in which single-dose pharmacokinetics of crizotinib or midazolam was characterized on Day-7, prior to initiation of continuous dosing in the first cycle (each cycle 28 days) of treatment in dose escalation cohorts and recommended phase 2 dose (RP2D) cohorts.
Groups:
- Low Dose Escalation Cohort: Crizotinib 50 mg QD: Participants received Crizotinib 50 milligram (mg) capsule or tablet orally once daily (QD) for up to 34 cycles (each cycle 28 days).
- Low Dose Escalation Cohort: Crizotinib 100 mg QD: Participants received Crizotinib 100 mg capsule or tablet orally QD for up to 34 cycles (each cycle 28 days) and 2 mg oral dose of Midazolam along with Crizotinib 100 mg on Cycle 2 Day 1 only. Participants who did not receive Crizotinib on Day -7, received single 2 mg oral dose of Midazolam on Day -7.
- Low Dose Escalation Cohort: Crizotinib 200 mg QD: Participants received Crizotinib 200 mg (2 capsules/tablet of 100 mg each) capsule/tablet orally QD for up to 34 cycles (each cycle 28 days).
- Low Dose Escalation Cohort: Crizotinib 200 mg BID: Participants received Crizotinib 200 mg (2 capsules/tablet of 100 mg each) capsule/tablet orally twice daily (BID) for up to 34 cycles (each cycle 28 days).
- Low Dose Escalation Cohort: Crizotinib 250 mg BID: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet BID for up to 34 cycles (each cycle 28 days).
- Low Dose Escalation Cohort: Crizotinib 300 mg BID: Participants received Crizotinib 300 mg (3 capsules/tablet of 100 mg each) capsule/tablet orally BID for up to 34 cycles (each cycle 28 days) and 2 mg oral dose of Midazolam along with Crizotinib 300 mg on Cycle 2 Day 1 only. Participants who did not receive Crizotinib on Day -7, received single 2 mg oral dose of Midazolam on Day -7.
- High Dose Escalation Cohort: Crizotinib 300 mg QD: Participants received Crizotinib 300 mg (3 capsules/tablet of 100 mg each) capsule/tablet QD for up to 7 cycles (each cycle 28 days).
- High Dose Escalation Cohort: Crizotinib 400 mg QD: Participants received Crizotinib 400 mg (4 capsules/tablet of 100 mg each) capsule/tablet QD for up to 7 cycles (each cycle 28 days).
- High Dose Escalation Cohort: Crizotinib 500 mg QD: Participants received Crizotinib 500 mg (5 capsules/tablet of 100 mg each) capsule/tablet QD for up to 7 cycles (each cycle 28 days).
- High Dose Escalation Cohort: Crizotinib 650 mg QD: Participants received Crizotinib 650 mg (6 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) for up to 7 cycles (each cycle 28 days).
- High Dose Escalation Cohort: Crizotinib 800 mg QD: Participants received Crizotinib 800 mg (8 capsules/tablet of 100 mg each) capsule/tablet QD for up to 7 cycles (each cycle 28 days).
- RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally twice daily (BID) with or without food for up to 105 cycles (each cycle 28 days).
- RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally twice daily (BID) with or without food for up to 55 cycles (each cycle 28 days).
- RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally twice daily (BID) with or without food for up to 101 cycles (each cycle 28 days).
- RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) with or without food for up to 70 cycles (each cycle 21 days).
- RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally BID with or without food for up to 70 cycles (each cycle 21 days).
- RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) with or without food for up to 133 cycles (each cycle 28 days).
- RP2D Cohort: Enriched Other: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally twice daily (BID) with or without food for up to 54 cycles (each cycle 28 days).
- RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg +Itraconazole: Participants received with or without food Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet QD from Cycle 1Day1 to Cycle 2 Day1 thereafter 250 mg BID from Cycle 2 Day 2 up to 58 cycles (each cycle 28 days). Participants also received Itraconazole 200 mg QD from Cycle 1 Day 1 to Cycle 1 Day 16.
- RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) with or without food from Cycle 1 Day 1 up to 13 cycles (each cycle 28 days). Participants also received commercially available Rifampin 650 mg QD from Cycle 1 Day 16 to Cycle 2 Day 1 (14 days) either one hour before or 2 hours after food.
- RP2D Cohort: Midazolam Interaction: Crizotinib 250 mg +Midazolam: Participants received Crizotinib 250 mg tablet/capsule (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) orally BID with or without food from Day 1 Cycle 1 up to 133 cycles (each cycle 28 days). Participants also received single 2 mg oral dose of Midazolam on Day -7 and another single 2-mg oral dose of Midazolam concurrently with Crizotinib on Cycle 2 Day 1
Period: Overall Study
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: Enriched Other: Crizotinib 250 mg | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg +Itraconazole | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin | RP2D Cohort: Midazolam Interaction: Crizotinib 250 mg +Midazolam
Started | 3 | 4 | 9 | 7 | 9 | 6 | 7 | 5 | 3 | 6 | 11 | 53 | 85 | 41 | 48 | 19 | 154 | 67 | 21 | 18 | 14
Treated | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9 | 53 | 85 | 41 | 48 | 18 | 154 | 66 | 18 | 18 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 9 | 7 | 9 | 6 | 7 | 5 | 3 | 6 | 11 | 53 | 85 | 41 | 48 | 19 | 154 | 67 | 21 | 18 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 8 | 6 | 4 | 1 | 14 | 9 | 2 | 3 | 1
Not completed — Progressive Disease | 2 | 2 | 5 | 4 | 6 | 4 | 6 | 3 | 0 | 5 | 2 | 25 | 29 | 26 | 21 | 12 | 94 | 42 | 4 | 9 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 8 | 15 | 0 | 3 | 0 | 7 | 1 | 2 | 2 | 0
Not completed — Other | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 19 | 24 | 7 | 11 | 3 | 28 | 12 | 10 | 4 | 2
Not completed — Randomized not treated | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 7 | 2 | 8 | 2 | 11 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn Due to Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis (SA) set included all enrolled participants who received at least one dose of Crizotinib on Cycle 1 Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: Enriched Other: Crizotinib 250 mg | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg +Itraconazole | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin | RP2D Cohort: Midazolam Interaction: Crizotinib 250 mg +Midazolam | Total
Number analyzed (Participants) | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9 | 53 | 85 | 41 | 48 | 18 | 154 | 66 | 18 | 18 | 12 | 578
Age, Customized [Count of Participants; unit: Participants]
  less than 65 years | 3 | 4 | 5 | 5 | 8 | 6 | 3 | 5 | 3 | 6 | 5 | 23 | 18 | 20 | 30 | 12 | 131 | 51 | 9 | 12 | 9 | 368
  greater than or equals to 65 years | 0 | 0 | 3 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 30 | 67 | 21 | 18 | 6 | 23 | 15 | 9 | 6 | 3 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 3 | 4 | 2 | 3 | 5 | 0 | 1 | 3 | 30 | 48 | 19 | 24 | 8 | 80 | 25 | 11 | 9 | 8 | 289
  Male | 0 | 3 | 6 | 4 | 4 | 4 | 3 | 0 | 3 | 5 | 6 | 23 | 37 | 22 | 24 | 10 | 74 | 41 | 7 | 9 | 4 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 7 | 6 | 8 | 6 | 6 | 4 | 2 | 5 | 8 | 30 | 60 | 38 | 35 | 11 | 98 | 49 | 13 | 16 | 11 | 418
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 3 | 5 | 4 | 3 | 2 | 0 | 27
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 21 | 15 | 1 | 9 | 2 | 43 | 9 | 0 | 0 | 0 | 102
  Other | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8 | 0 | 3 | 2 | 8 | 4 | 2 | 0 | 1 | 31

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Cohort: Maximum Tolerated Dose (MTD) of Crizotinib
Description: MTD: Dose level at which at most 1 of 6 participants experienced DLT within and including 28 days of treatment (during Cycle 1 [1 cycle=28 days]) with next higher dose having at least 2/3 or 2/6 participants experiencing a DLT. DLT was defined as any of following: Hematologic toxicities- 1) prolonged grade 4 neutropenia for >7 days. 2) Febrile neutropenia: grade 4 neutropenia with fever greater than (>) 38.5 degree Celsius, both sustained over a 24 hour period (3) neutropenic infection: greater than or equal to (>=) Grade 3 neutropenia with Grade >=3 infection. (4) Grade >=3 thrombocytopenia with bleeding/grade 4 lasting >=7 days. Other non-hematologic toxicity included: Grade 3/4 toxicities (except for alopecia, Grade 3/4 hypophosphatemia, grade 3 hypertension with controlled blood pressure [less than (<) 140/90 millimeter of mercury, and Grade 3/4 hyperuricemia without signs and symptoms of gout). Nausea, vomiting/diarrhea must persist at grade 3/4 despite maximal medical therapy.
Time Frame: Cycle 1 (28 days)
Population: as for baseline characteristics
Measure: Number; unit: milligram
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD
Number analyzed (Participants) | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9
milligram | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250

2. Primary Outcome: Dose-Escalation Cohort: Recommended Phase 2 Dose (RP2D) of Crizotinib
Description: RP2D was defined as a dose below or equal to MTD, at which crizotinib was unlikely to cause a significant inhibition of CYP3A4 activity.
Time Frame: Cycle 1 (28 days)
Population: as for baseline characteristics
Measure: Number; unit: milligram
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD
Number analyzed (Participants) | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9
milligram | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250

3. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Crizotinib on Day -7
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) extrapolated to infinite time (0-inf).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9, 24, 48 and any two time points (72, 96, 120 and 144 hours) post-dose on Day -7
Population: Pharmacokinetic (PK) parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. "Overall number of participants analyzed (N)" signifies participants evaluable for this outcome measure (OM). Data for this OM was planned to be collected for individual arms of low and high dose escalation and combined RP2D Cohort excluding "Low Dose Escalation Cohort: Crizotinib 100 mg QD" arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Groups:
- RP2D Cohort: Crizotinib 250 mg: Participants received Crizotinib 250 mg tablet/capsule (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) orally BID up to 124 months.
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 7 | 2 | 8 | 1 | 5 | 5 | 2 | 6 | 8 | 29
nanogram*hour per milliliter | 274.43 (22) | 1378.05 (144) | 946.93 (38) | 1817.35 (34) | 2320.00 | 3457 (42) | 3078 (119) | 2107 (53) | 3979 (39) | 7547 (76) | 2489.39 (53)

4. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib on Day -7
Description: Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau), where dosing interval is 12 hours for BID dose and 24 hours for QD dose.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9, 24, 48 and any two time points (72, 96, 120 and 144 hours) post-dose on Day -7
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be reported for individual arms of low and high dose escalation and combined RP2D Cohort excluding "Low Dose Escalation Cohort: Crizotinib 100 mg QD" arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 8 | 5 | 9 | 1 | 6 | 5 | 3 | 6 | 8 | 46
nanogram*hour per milliliter | 137.40 (8) | 658.64 (136) | 338.39 (50) | 558.01 (33) | 863.00 | 1731 (51) | 1377 (114) | 1300 (61) | 1906 (39) | 3423 (57) | 741.50 (45)

5. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib on Cycle 1 Day 1
Description: as for outcome 4
Time Frame: Pre-dose, 2, 4 and 6 hours post dose on Cycle 1 Day 1
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be collected for low dose escalation cohort (excluding Crizotinib 50 mg QD, Crizotinib 200 mg QD and Crizotinib 250 mg BID arms) and combined RP2D cohort and was not planned to be collected for high dose escalation cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 4 | 2 | 5 | 88
nanogram*hour per milliliter | 457.55 (32) | 383.98 (10) | 763.71 (57) | 663.39 (56)

6. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib on Cycle 1 Day 15
Description: as for outcome 4
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 1 Day 15
Population: The PK parameter analysis population included all participants treated (including Day -7 dose) who have at least 1 of the PK parameters of interest for Crizotinib. Here, "Overall number of participants analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measures was planned to be collected for individual arms of dose escalation cohorts and combined RP2D Cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 4 | 8 | 4 | 5 | 4 | 6 | 2 | 3 | 5 | 3 | 19
nanogram*hour per milliliter | 206.13 (76) | 1086.99 (34) | 2047.13 (45) | 1780.21 (69) | 3083.93 (31) | 4066.67 (53) | 4375 (34) | 3385 (24) | 6655 (4) | 6362 (37) | 10480 (76) | 3879.56 (45)

7. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib on Cycle 2 Day 1
Description: as for outcome 4
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 2 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 2 | 5 | 3 | 2 | 4 | 2 | 16
nanogram*hour per milliliter | 425.90 (49) | 1595.58 (30) | 1719.30 (68) | 2255.70 (14) | 3054.45 (29) | 3644.72 (17) | 4815 (23) | 3839 (65) | 6330 (64) | 7273 (48) | 8733 (63) | 4163.77 (40)

8. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Trough Concentration (Ctrough) of Crizotinib Cycle 1 Day 15
Description: Ctrough refers to plasma concentration of Crizotinib observed just before treatment administration.
Time Frame: Pre-dose on Cycle 1 Day 15
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be collected for individual arms of low dose escalation and combined RP2D Cohort and not planned to be collected for high dose escalation cohort".
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 4 | 8 | 3 | 5 | 4 | 24
nanogram per milliliter | 7.29 (42) | 32.61 (36) | 48.18 (58) | 126.76 (97) | 232.59 (33) | 307.83 (59) | 280.43 (75)

9. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Trough Concentration (Ctrough) of Crizotinib on Cycle 2 Day 1
Description: Ctrough refers to plasma concentration of Crizotinib observed just before treatment administration.
Time Frame: Pre-dose on Cycle 2 Day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 3 | 18
nanogram per milliliter | 12.68 (94) | 31.91 (34) | 54.04 (85) | 157.24 (17) | 232.45 (32) | 329.50 (40) | 312.99 (55)

10. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib on Day -7
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9, 24, 48 and any two time points (72, 96, 120 and 144 hours) post-dose on Day -7
Population: PK parameter analysis population set. "N"=participants evaluable for this outcome measure. Data for this OM was planned to be collected for dose escalation cohorts (both low and high) and combined RP2D Cohort excluding "Low Dose Escalation Cohort: Crizotinib 100 mg QD" cohort arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 8 | 5 | 9 | 1 | 6 | 5 | 3 | 6 | 8 | 46
nanogram per milliliter | 24.19 (36) | 67.64 (106) | 55.73 (45) | 87.02 (34) | 130.00 | 184.7 (65) | 115.9 (85) | 146.6 (31) | 154.3 (30) | 270.9 (47) | 108.40 (42)

11. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib on Cycle 1 Day 1
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: Pre-dose, 2, 4 and 6 hours post dose on Cycle 1 Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 4 | 2 | 5 | 98
nanogram per milliliter | 54.89 (53) | 64.14 (2) | 114.09 (48) | 98.86 (55)

12. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib on Cycle 1 Day 15
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 1 Day 15
Population: The PK parameter analysis population included all participants treated (including Day -7 dose) who have at least 1 of the PK parameters of interest for Crizotinib. Here, "Overall number of participants analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measures was planned to be collected for individual arms of dose escalation cohorts (both low and high) and combined RP2D Cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 4 | 8 | 4 | 5 | 4 | 6 | 3 | 3 | 5 | 4 | 24
nanogram per milliliter | 24.44 (68) | 85.66 (66) | 149.06 (29) | 188.84 (56) | 326.51 (24) | 420.15 (46) | 315.2 (50) | 215.5 (26) | 395.3 (16) | 379.2 (28) | 671.3 (76) | 411.11 (51)

13. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib on Cycle 2 Day 1
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 2 Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 5 | 3 | 6 | 3 | 2 | 4 | 2 | 18
nanogram per milliliter | 47.99 (23) | 133.69 (48) | 146.26 (38) | 238.84 (12) | 327.94 (25) | 474.68 (43) | 275.0 (28) | 248.2 (60) | 327.9 (47) | 419.8 (36) | 700.0 (37) | 477.85 (44)

14. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crizotinib on Day -7
Description: Tmax was defined as the time to reach the observed maximum plasma concentration (Cmax).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9, 24, 48 and any two time points (72, 96, 120 and 144 hours) post-dose on Day -7
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be collected for individual arms of low and high dose escalation cohorts (excluding 'Low Dose Escalation Cohort: Crizotinib 100 mg QD' arm) and combined RP2D.
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 8 | 5 | 9 | 1 | 6 | 5 | 3 | 6 | 8 | 46
hour | 2.00 [1.75 to 4.08] | 4.09 [1.08 to 6.00] | 4.00 [4.00 to 4.08] | 4.00 [1.00 to 8.95] | 2.02 [2.02 to 2.02] | 4.00 [2.00 to 6.00] | 2.15 [1.00 to 6.00] | 4.00 [2.00 to 8.00] | 4.00 [1.98 to 6.00] | 4.99 [2.15 to 6.13] | 4.00 [2.00 to 9.33]

15. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crizotinib on Cycle 1 Day 1
Description: Tmax was defined as the time to reach the observed maximum plasma concentration (Cmax).
Time Frame: Pre-dose, 2, 4 and 6 hours post dose on Cycle 1 Day 1
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be collected for low dose escalation cohorts (excluding Crizotinib 50 mg QD, Crizotinib 200 mg QD and Crizotinib 250 mg BID arms) and combined RP2D cohort and was not planned to be collected for high dose escalation cohort.
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 4 | 2 | 5 | 98
hour | 2.52 [1.00 to 4.02] | 4.00 [4.00 to 4.00] | 4.00 [2.05 to 8.02] | 4.05 [1.00 to 9.08]

16. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crizotinib on Cycle 1 Day 15
Description: Tmax was defined as the time to reach the observed maximum plasma concentration (Cmax).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 4 | 8 | 4 | 5 | 4 | 6 | 3 | 3 | 5 | 4 | 24
hour | 2.00 [1.00 to 4.00] | 2.51 [0.00 to 6.08] | 4.07 [1.00 to 6.00] | 5.01 [2.08 to 8.03] | 4.00 [0.97 to 6.07] | 4.99 [3.98 to 6.22] | 5.13 [1.93 to 7.88] | 5.17 [0.933 to 6.00] | 4.00 [4.00 to 9.00] | 5.98 [4.00 to 6.00] | 5.03 [4.00 to 6.03] | 4.00 [0.00 to 9.03]

17. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crizotinib Cycle 2 Day 1
Description: Tmax was defined as the time to reach the observed maximum plasma concentration (Cmax).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 2 Day 1
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 3 | 6 | 3 | 2 | 4 | 2 | 18
hour | 1.02 [1.00 to 4.00] | 3.98 [2.00 to 4.02] | 4.00 [2.00 to 4.17] | 4.00 [3.95 to 4.00] | 4.00 [4.00 to 6.00] | 4.05 [3.98 to 9.00] | 3.00 [1.00 to 5.95] | 4.00 [2.08 to 6.00] | 7.59 [6.18 to 9.00] | 4.30 [4.00 to 9.00] | 5.00 [4.00 to 6.00] | 4.00 [0.00 to 9.02]

18. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Plasma Decay Half-Life (t1/2) of Crizotinib on Day -7
Description: Plasma decay half-life is the time measured for the plasma concentration of Crizotinib to decrease by one half.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 9, 24, 48 and any two time points (72, 96, 120 and 144 hours) post-dose on Day -7
Population: PK parameter analysis population included all participants treated (including Day -7 dose) who had at least 1 of the PK parameters of interest for Crizotinib. Here, "N" signifies participants evaluable for this OM. Data for this OM was planned to be collected for individual arms of low and high dose escalation cohort and combined RP2D cohort excluding "Low Dose Escalation Cohort: Crizotinib 100 mg QD" arm.
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3 | 7 | 2 | 8 | 1 | 5 | 5 | 2 | 6 | 8 | 31
hour | 48.20 [45.50 to 56.80] | 46.70 [30.40 to 67.20] | 52.60 [51.70 to 53.50] | 47.35 [36.80 to 57.70] | 45.70 [45.70 to 45.70] | 43.33 [35.4 to 52.3] | 49.06 [33.2 to 79.3] | 46.36 [43.0 to 49.8] | 42.17 [28.3 to 53.8] | 38.78 [30.9 to 55.3] | 43.20 [27.10 to 63.40]

19. Primary Outcome: Dose-Escalation and Recommended Phase 2 Dose (RP2D) Cohort: Number of Participants With Treatment Emergent Adverse Events (TEAES) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. AEs included both serious and all non-serious adverse events. TEAEs were those with initial onset or increasing in severity on or after the first dose of investigational product administration.
Time Frame: up to 189 Months
Population: SA set included all enrolled participants who received at least one dose of Crizotinib on Cycle 1 Day 1.
Measure: Count of Participants; unit: Participants
Groups:
- RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet orally twice daily (BID) with or without food for up to 105 cycles (each cycle 28 days)
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: Enriched Other: Crizotinib 250 mg | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg +Itraconazole | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin | RP2D Cohort: Midazolam Interaction: Crizotinib 250 mg +Midazolam
Number analyzed (Participants) | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9 | 53 | 85 | 41 | 48 | 18 | 154 | 66 | 18 | 18 | 12
Participants
  AEs | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 4 | 3 | 6 | 9 | 53 | 85 | 41 | 47 | 18 | 154 | 66 | 18 | 18 | 12
  SAEs | 0 | 0 | 1 | 2 | 4 | 2 | 2 | 2 | 1 | 2 | 4 | 24 | 54 | 25 | 22 | 9 | 75 | 29 | 7 | 6 | 6

20. Primary Outcome: Dose-Escalation Cohort: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Dose-limiting toxicity (DLT) was defined as any of the following: Hematologic- prolonged grade 4 neutropenia for >7 days. Febrile neutropenia, defined as grade 4 neutropenia with fever greater than (>)38.5 degree Celsius, both sustained over a 24 hour period, neutropenic infection: greater than or equal to (>=)Grade 3 neutropenia with Grade >=3 infection. Grade >=3 thrombocytopenia with bleeding or grade 4 lasting >=7 days Lymphopenia was not considered a DLT unless accompanied by infection. Other non-hematologic toxicity: Grade 3 or 4 toxicities (except for alopecia, Grade 3/4 hypophosphatemia, grade 3 hypertension with controlled blood pressure [less than (<) 140/90], and Grade 3/4 hyperuricemia without signs and symptoms of gout). Nausea, vomiting or diarrhea must persist at grade 3 or 4 despite maximal medical therapy.
Time Frame: Cycle 1 (28 days)
Population: SA set included all enrolled participants who received at least one dose of Crizotinib on Cycle 1 Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD
Number analyzed (Participants) | 3 | 4 | 8 | 7 | 8 | 6 | 6 | 5 | 3 | 6 | 9
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Midazolam Interaction Cohort: Maximum Observed Plasma Concentration (Cmax) of Midazolam When Taken Alone or Taken With Crizotinib
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 9, and 24 hours post dose on Day -7 (midazolam alone arm), pre-dose, 0.5, 1, 2, 4, 6, 8, 9, and 24 hours post dose on Cycle 2 Day 1 (midazolam with crizotinib arm)
Population: The PK concentration population of midazolam included all participants treated with midazolam (including Day -7 dose) who have at least 1 concentration of midazolam.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Groups:
- Low Dose Escalation Cohort: Crizotinib 100 mg QD (Midazolam Alone): Participants who did not receive Crizotinib on Day -7, received single 2 mg oral dose of Midazolam on Day -7.
- Low Dose Escalation Cohort: Crizotinib 100 mg QD + Midazolam: Participants received Crizotinib 100 mg capsule or tablet orally QD along with single 2 mg oral dose of Midazolam on Cycle 2 Day 1.
- Low Dose Escalation Cohort: Crizotinib 300 mg BID (Midazolam Alone): Participants who did not receive Crizotinib 300 mg (3 capsules/tablet of 100 mg each) capsule/tablet BID on Day -7, received single 2 mg oral dose of Midazolam on Day -7.
- Low Dose Escalation Cohort: Crizotinib 300 mg BID + Midazolam: Participants received Crizotinib 300 mg (3 capsules/tablet of 100 mg each) capsule/tablet orally BID along with 2 mg oral dose of Midazolam on Cycle 2 Day 1.
- RP2D Cohort: Crizotinib 250 mg (Midazolam Alone): Participants who did not receive Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet on Day -7, received single 2 mg oral dose of Midazolam on Day -7.
- RP2D Cohort: Crizotinib 250 mg + Midazolam: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) BID along with single 2 mg oral dose of Midazolam on Cycle 2 Day 1.
Arm/Group | Low Dose Escalation Cohort: Crizotinib 100 mg QD (Midazolam Alone) | Low Dose Escalation Cohort: Crizotinib 100 mg QD + Midazolam | Low Dose Escalation Cohort: Crizotinib 300 mg BID (Midazolam Alone) | Low Dose Escalation Cohort: Crizotinib 300 mg BID + Midazolam | RP2D Cohort: Crizotinib 250 mg (Midazolam Alone) | RP2D Cohort: Crizotinib 250 mg + Midazolam
Number analyzed (Participants) | 4 | 3 | 5 | 2 | 14 | 8
nanogram per milliliter | 14.98 (19) | 19.26 (38) | 13.65 (10) | 32.62 (40) | 12.78 (41) | 25.37 (67)
Statistical Analysis 1: Comparison: Low Dose Escalation Cohort: Crizotinib 100 mg QD (Midazolam Alone) vs Low Dose Escalation Cohort: Crizotinib 100 mg QD + Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 131.72, 90% CI 2-sided [96.59 to 179.63]
Statistical Analysis 2: Comparison: Low Dose Escalation Cohort: Crizotinib 300 mg BID (Midazolam Alone) vs Low Dose Escalation Cohort: Crizotinib 300 mg BID + Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 239.03, 90% CI 2-sided [172.14 to 331.93]
Statistical Analysis 3: Comparison: RP2D Cohort: Crizotinib 250 mg (Midazolam Alone) vs RP2D Cohort: Crizotinib 250 mg + Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 201.56, 90% CI 2-sided [139.33 to 291.58]

22. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Midazolam When Taken Alone or Taken With Crizotinib
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Groups:
- RP2D Cohort: Crizotinib 250 mg +Midazolam: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) BID along with single 2 mg oral dose of Midazolam on Cycle 2 Day 1.
Arm/Group | Low Dose Escalation Cohort: Crizotinib 100 mg QD (Midazolam Alone) | Low Dose Escalation Cohort: Crizotinib 100 mg QD + Midazolam | Low Dose Escalation Cohort: Crizotinib 300 mg BID (Midazolam Alone) | Low Dose Escalation Cohort: Crizotinib 300 mg BID + Midazolam | RP2D Cohort: Crizotinib 250 mg (Midazolam Alone) | RP2D Cohort: Crizotinib 250 mg +Midazolam
Number analyzed (Participants) | 4 | 3 | 5 | 2 | 14 | 8
nanogram*hour per milliliter | 41.77 (27) | 90.78 (33) | 37.71 (38) | 151.45 (31) | 32.10 (36) | 112.78 (87)
Statistical Analysis 1: Comparison: Low Dose Escalation Cohort: Crizotinib 100 mg QD (Midazolam Alone) vs Low Dose Escalation Cohort: Crizotinib 100 mg QD + Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 216.19, 90% CI 2-sided [161.41 to 289.56]
Statistical Analysis 2: Comparison: Low Dose Escalation Cohort: Crizotinib 300 mg BID (Midazolam Alone) vs Low Dose Escalation Cohort: Crizotinib 300 mg BID + Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 350.00, 90% CI 2-sided [141.09 to 868.23]
Statistical Analysis 3: Comparison: RP2D Cohort: Crizotinib 250 mg (Midazolam Alone) vs RP2D Cohort: Crizotinib 250 mg +Midazolam; Test type: Superiority; Ratio of adjusted geometric means = 365.43, 90% CI 2-sided [263.22 to 507.31]

23. Primary Outcome: RP2D Cohort: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] of Crizotinib When Taken With Food
Description: AUC0-24 of Crizotinib was defined as the area under the free plasma concentration time curve from time 0 to 24 hours post-dose.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 9, and 24 hours post-dose on Day -7
Population: The food effect analysis set included all participants treated (including Day -7 dose) and in the RP2D cohort who had received a dose of crizotinib under fed conditions and for which at least 1 PK parameter of interest (Cmax or AUC) was available. Here, "Overall number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Groups:
- RP2D Cohort: Crizotinib 250 mg With Food: Participants who were enrolled in enriched RP2D cohort received single dose of Crizotinib 250 mg tablet/capsule (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) orally with food on Day -7.
Arm/Group | RP2D Cohort: Crizotinib 250 mg With Food
Number analyzed (Participants) | 8
nanogram*hour per milliliter | 1212.86 (46)

24. Primary Outcome: RP2D Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib When Taken With Food
Description: Cmax is defined as the observed maximum plasma concentration post drug administration.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 9, and 24 hours post-dose on Day -7
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | RP2D Cohort: Crizotinib 250 mg With Food
Number analyzed (Participants) | 11
nanogram per milliliter | 106.24 (51)

25. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib Alone and When Taken With Rifampin
Description: Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau).
Time Frame: pre-dose, 2, 4, 6, 8 and 10 hours on Cycle 1 Day 15 (Crizotinib alone arm) and Cycle 2 Day 1 (Crizotinib with Rifampin arm)
Population: PK parameter population was defined as all participants in the Rifampin interaction cohort safety population who satisfied following criteria for Cycle 1 Day 15 or Cycle 2 Day 1: a) had at least 1 of the primary PK parameters of Crizotinib (AUCtau and Cmax). b) received adequate dosing prior to PK sampling. Here, "Overall number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Groups:
- RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) with or without food from Cycle 1 Day 1 up to 13 cycles (each cycle 28 days).
- RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet twice daily (BID) form Cycle 1Day 1 up to 13 cycles (each cycle 28 days). Participants also received commercially available Rifampin 650 mg QD from Cycle 1 Day 16 to Cycle 2 Day 1 (14 days) either one hour before or 2 hours after a meal.
Arm/Group | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin
Number analyzed (Participants) | 10 | 7
nanogram*hour per milliliter | 3110 (49) | 509.6 (35)
Statistical Analysis 1: Comparison: RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone vs RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin; Test type: Superiority; Ratio of adjusted geometric mean = 15.57, 90% CI 2-sided [10.89 to 22.26]

26. Primary Outcome: Rifampin Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib Alone and When Taken With Rifampin
Time Frame: pre-dose, 2, 4, 6, 8 and 10 hours on Cycle 1 Day 15 (Crizotinib alone) and Cycle 2 Day 1 (Crizotinib with Rifampin)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin
Number analyzed (Participants) | 10 | 7
nanogram per milliliter | 326.4 (48) | 71.53 (49)
Statistical Analysis 1: Comparison: RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone vs RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin; Test type: Superiority; Ratio of adjusted geometric mean = 20.64, 90% CI 2-sided [14.59 to 29.18]

27. Primary Outcome: Rifampin Cohort: Ctrough of Crizotinib Alone and When Taken With Rifampin
Description: Ctrough refers to plasma concentration of Crizotinib observed just before treatment administration.
Time Frame: pre-dose on Cycle 1 Day 15 (Crizotinib alone arm) and Cycle 2 Day 1 (Crizotinib with Rifampin arm)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg Alone | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg With Rifampin
Number analyzed (Participants) | 9 | 7
nanogram per milliliter | 251.7 (46) | 26.67 (50)

28. Primary Outcome: Itraconazole Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib When Taken Alone and When Taken With Itraconazole
Description: Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau), where dosing interval is 24 hours.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 9 and 24 hours post dose on Cycle 1 Day 15 (Crizotinib with itraconazole) and Cycle 2 Day 1 (itraconazole alone)
Population: PK parameter evaluable population included participants who had at least 1 of the PK parameters of Crizotinib (AUCtau or Cmax) and had received 10 consecutive doses of both Crizotinib 250 mg QD and itraconazole 200 mg QD immediately prior to end of Crizotinib 250 mg + Itraconazole treatment as well as 10 consecutive doses of Crizotinib 250 mg QD prior to end of Crizotinib 250 mg + Itraconazole treatment. Overall number of participants analyzed =participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Groups:
- RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone: Participants received with or without food Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet QD from Cycle 1Day1 to Cycle 2 Day1 thereafter 250 mg BID from Cycle 2 Day 2 up to 58 cycles (each cycle 28 days).
- Itraconazole Interaction Cohort: Crizotinib 250 mg + Itraconazole: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet QD from Cycle 1Day1 to Cycle 2 Day1 thereafter 250 mg BID from Cycle 2 Day 2 up to 58 cycles (each cycle 28 days). Participants also received Itraconazole 200 mg QD from Cycle 1 Day 1 to Cycle 1 Day 16. (each cycle 28 days).
Arm/Group | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone | Itraconazole Interaction Cohort: Crizotinib 250 mg + Itraconazole
Number analyzed (Participants) | 10 | 10
nanogram*hour per milliliter | 4102 (31) | 6665 (16)
Statistical Analysis 1: Comparison: RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone vs Itraconazole Interaction Cohort: Crizotinib 250 mg + Itraconazole; Test type: Superiority; Ratio of adjusted geometric means = 157.40, 90% CI 2-sided [136.89 to 180.97]

29. Primary Outcome: Itraconazole Cohort: Maximum Observed Plasma Concentration (Cmax) of Crizotinib When Taken Alone and When Taken With Itraconazole
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Groups:
- RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg With Itraconazole: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet QD from Cycle 1Day1 to Cycle 2 Day1 thereafter 250 mg BID from Cycle 2 Day 2 up to 58 cycles (each cycle 28 days). Participants also received Itraconazole 200 mg QD from Cycle 1 Day 1 to Cycle 1 Day 16. (each cycle 28 days).
Arm/Group | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg With Itraconazole
Number analyzed (Participants) | 10 | 10
nanogram per milliliter | 259.9 (23) | 353.2 (14)
Statistical Analysis 1: Comparison: RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone vs RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg With Itraconazole; Test type: Superiority; Ratio of adjusted geometric means = 132.81, 90% CI 2-sided [119.10 to 148.10]

30. Primary Outcome: Itraconazole Cohort: Trough Plasma Concentration (Ctrough) of Crizotinib When Taken Alone and When Taken With Itraconazole
Description: Ctrough refers to plasma concentration of Crizotinib observed just before treatment administration.
Time Frame: pre-dose on Cycle 1 Day 15 (crizotinib with itraconazole) and Cycle 2 Day 1 (itraconazole alone)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg Alone | RP2D Cohort: Itraconazole Interaction: Crizotinib 250 mg With Itraconazole
Number analyzed (Participants) | 7 | 9
nanogram per milliliter | 136.0 (36) | 214.0 (30)

31. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Percentage of Participants With Objective Response (OR)
Description: ORR was defined as participants with a best overall response of complete response (CR) or partial response (PR) divided by the total number of evaluable participants per RECIST version 1.0 (RECIST1.1 for ALK-negative NSCLC cohort 1 and ALK-negative NSCLC cohort 2). CR: Disappearance of all target and non-target lesions, normalization of tumor marker levels, and no appearance of new lesions indicated complete response. PR: At least a 30% decrease in the sum of the longest diameters of target lesions (taking as reference the baseline sum), without progression of non-target lesions and no appearance of new lesions indicated partial response.
Time Frame: Baseline up to 172 months
Population: Response-evaluable population was defined as all participants in the SA set who had an adequate baseline disease assessment and had met 1 of the following 2 criteria: a) Had at least one post-baseline disease assessment b) withdrew from the trial or experienced progression/death at any time on study. Here, "Overall number of participants Analyzed" signifies number of participants evaluable for this outcome measure. Data was planned to be analyzed for reported arms only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: Enriched Other: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 65 | 38 | 18 | 116 | 66
percentage of participants | 71.7 [57.7 to 83.2] | 32.3 [21.2 to 45.1] | 31.6 [17.5 to 48.7] | 19.0 [5.4 to 41.9] | 61.2 [51.7 to 70.1] | 8.3 [0.2 to 38.5]

32. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Duration of Response (DOR)
Description: Duration of response (DoR) was the time from first documentation of PR or CR to date of first documentation of progressive disease (PD) or death due to any cause. PR: At least a 30% decrease in the sum of the longest diameters of target lesions (taking as reference the baseline sum), without progression of non-target lesions and no appearance of new lesions indicated partial response. CR: Disappearance of all target and non-target lesions, normalization of tumor marker levels, and no appearance of new lesions indicated complete response. PD: >=20% increase in the sum of the longest diameter of target lesions taking as references the smallest sum longest diameter recorded since the treatment started, unequivocal progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: From first documentation of response to date of PD or death due to any cause (up to 172 months)
Population: Response-evaluable population was defined as all participants in the SA set who had an adequate baseline disease assessment and had met 1 of the following 2 criteria: a) Had at least one post-baseline disease assessment b) withdrew from the trial or experienced progression/death at any time on study. Here, "Overall number of participants analyzed" signifies number of participants who were objective responders. Data was planned to be analyzed for reported arms only.
Measure: Median (Full Range); unit: Weeks
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 38 | 33 | 12 | 71
Weeks | 14.5 [2.8 to 45.4] | 6.8 [2.8 to 13.4] | 5.2 [3.8 to 12.2] | 26.2 [8.1 to 72.9]

33. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Time to Response (TTR)
Description: TTR: time between first dose until first documented response of PR or CR. PR: At least a 30% decrease in the sum of the longest diameters of target lesions (taking as reference the baseline sum), without progression of non-target lesions and no appearance of new lesions indicated partial response. CR: Disappearance of all target and non-target lesions, normalization of tumor marker levels, and no appearance of new lesions indicated complete response.
Time Frame: From first dose until first documented response of PR or CR (up to 172 months)
Population: as for outcome 32
Measure: Median (Full Range); unit: Weeks
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 38 | 33 | 12 | 71
Weeks | 7.9 [4.3 to 103.6] | 7.6 [3.7 to 47.3] | 8.0 [7.1 to 23.6] | 7.7 [4.3 to 39.6]

34. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Percentage of Participants With Disease Control at Week 8
Description: Disease control was defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD) per RECIST version 1.0 (RECIST1.1 for ALK-negative NSCLC cohort 1 and ALK-negative NSCLC cohort 2). PR: At least a 30% decrease in the sum of the longest diameters of target lesions (taking as reference the baseline sum), without progression of non-target lesions and no appearance of new lesions indicated partial response. CR: Disappearance of all target and non-target lesions, normalization of tumor marker levels, and no appearance of new lesions indicated complete response. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Week 8
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 116 | 18
percentage of participants | 86.8 [74.7 to 94.5] | 71.8 [61.0 to 81.0] | 79.3 [70.8 to 86.3] | 47.6 [25.7 to 70.2]

35. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Percentage of Participants With Disease Control at Week 16
Description: as for outcome 34
Time Frame: Week 16
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 116 | 18
percentage of participants | 79.2 [65.9 to 89.2] | 51.8 [40.7 to 62.7] | 67.2 [57.9 to 75.7] | 42.9 [21.8 to 66.0]

36. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was the time from randomization date to date of first documentation of PD or death due to any cause RECIST version 1.0 (RECIST1.1 for ALK-negative NSCLC cohort 1 and ALK-negative NSCLC cohort 2). PD: >=20% increase in the sum of the longest diameter of target lesions taking as references the smallest sum longest diameter recorded since the treatment started, unequivocal progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: From randomization until PD or death, whichever occurred first (up to 172 months)
Population: SA set included all enrolled participants who received at least one dose of Crizotinib on Cycle 1 Day 1. Here, "Overall number of participants analyzed" signifies number of participants evaluable for this outcome measure. Data was planned to be analyzed for reported arms only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 41 | 119
Months | 19.3 [15.2 to 39.1] | 7.6 [5.6 to 9.1] | 4.0 [1.9 to 6.9] | 10.0 [8.2 to 14.7]

37. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Probability of Being Event Free at Month 6
Description: Probability of being event free (event defined as PD or death due to any cause) at 6 months after the first dose of crizotinib was reported. PD: >=20% increase in the sum of the longest diameter of target lesions taking as references the smallest sum longest diameter recorded since the treatment started, unequivocal progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: From randomization to 6 months
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: Probability of being event-free
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 41 | 119
Probability of being event-free | 76.9 [62.8 to 86.1] | 57.5 [45.3 to 68.0] | 39.0 [22.8 to 54.9] | 71.9 [61.8 to 79.7]

38. Primary Outcome: Recommended Phase 2 Dose (RP2D) Cohort: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization date to the date of death (up to 172 Months)
Population: as for outcome 36
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 41 | 119
Months | 51.4 [29.3 to NA] — Upper limit of 95% CI could not be estimable due to low number of participants with events. | 20.0 [13.2 to 25.7] | 10.1 [7.1 to 12.9] | NA [NA to NA] — Median and 95% CI could not be estimable due to low number of participants with events.

39. Primary Outcome: Probability of Participant Survival at Month 6
Description: Probability of survival was defined as the probability of being alive at Month 6.
Time Frame: Month 6
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: Probability of participants survival
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 41 | 119
Probability of participants survival | 90.5 [78.7 to 95.9] | 86.7 [77.3 to 92.4] | 67.8 [51.1 to 79.9] | 90.0 [82.7 to 94.4]

40. Primary Outcome: Probability of Participant Survival at Month 12
Description: Probability of survival was defined as the probability of being alive at Month 12.
Time Frame: Month 12
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: probability of participants survival
Arm/Group | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg
Number analyzed (Participants) | 53 | 85 | 41 | 119
probability of participants survival | 78.8 [65.0 to 87.7] | 66.0 [54.0 to 75.5] | 37.1 [22.4 to 51.8] | 80.5 [70.9 to 87.2]

41. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 1 Day 15
Description: Geometric mean of ratio (Cycle1Day15/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts.
Time Frame: Baseline, Cycle 1 Day 15
Population: Hypogonadism test evaluable population: Male participants who had completed screening, had received at least 1 dose of crizotinib on Cycle 1 Day 1, had at least 1 post baseline visit data for at least total testosterone, free testosterone, SHBG and included male participants of MET amplification and enriched other Cohort following approval of protocol amendment number 21. "N" =participants evaluable for this OM and 'number analyzed' =participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 28
Ratio
  Testosterone: number analyzed (Participants) | 22
  Testosterone | 0.46 [0.34 to 0.62]
  Estradiol: number analyzed (Participants) | 19
  Estradiol | 0.53 [0.42 to 0.66]
  Prolactin: number analyzed (Participants) | 22
  Prolactin | 1.19 [0.91 to 1.55]
  Luteinizing Hormone (LH) Serum: number analyzed (Participants) | 22
  Luteinizing Hormone (LH) Serum | 0.58 [0.47 to 0.73]
  Follicle Stimulating Hormone: number analyzed (Participants) | 22
  Follicle Stimulating Hormone | 0.77 [0.66 to 0.91]
  Free Testosterone: number analyzed (Participants) | 22
  Free Testosterone | 0.96 [0.66 to 1.40]
  Sex Hormone Binding Globulin | 0.36 [0.32 to 0.41]
  Dihydroepiandrosterone Sulfate: number analyzed (Participants) | 21
  Dihydroepiandrosterone Sulfate | 0.97 [0.85 to 1.11]

42. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 2 Day 1
Description: Geometric mean of ratio (Cycle 2 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts.
Time Frame: Baseline, Cycle 2 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 25
Ratio
  Testosterone: number analyzed (Participants) | 24
  Testosterone | 0.47 [0.38 to 0.58]
  Estradiol: number analyzed (Participants) | 22
  Estradiol | 0.72 [0.56 to 0.93]
  Prolactin | 0.89 [0.71 to 1.12]
  LH Serum: number analyzed (Participants) | 23
  LH Serum | 0.42 [0.26 to 0.70]
  Follicle Stimulating Hormone: number analyzed (Participants) | 23
  Follicle Stimulating Hormone | 0.69 [0.48 to 1.00]
  Free Testosterone: number analyzed (Participants) | 24
  Free Testosterone | 1.31 [0.97 to 1.77]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 17
  Sex Hormone Binding Globulin | 0.24 [0.18 to 0.31]
  Dihydroepiandrosterone Sulfate | 0.85 [0.75 to 0.96]

43. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 4 Day 1
Description: Geometric mean of ratio (Cycle 4 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts.
Time Frame: Baseline, Cycle 4 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 10
Ratio
  Testosterone | 0.48 [0.27 to 0.84]
  Estradiol: number analyzed (Participants) | 8
  Estradiol | 0.66 [0.49 to 0.89]
  Prolactin | 0.84 [0.55 to 1.28]
  LH Serum | 0.75 [0.57 to 1.00]
  Follicle Stimulating Hormone | 0.88 [0.68 to 1.15]
  Free Testosterone | 1.63 [0.88 to 3.01]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 8
  Sex Hormone Binding Globulin | 0.22 [0.18 to 0.28]
  Dihydroepiandrosterone Sulfate | 0.81 [0.69 to 0.97]

44. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 6 Day 1
Description: Geometric mean of ratio (Cycle 6 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts.
Time Frame: Baseline, Cycle 6 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 10
Ratio
  Testosterone | 0.49 [0.24 to 1.01]
  Estradiol: number analyzed (Participants) | 8
  Estradiol | 0.75 [0.58 to 0.97]
  Prolactin | 0.69 [0.48 to 1.00]
  LH Serum | 0.78 [0.60 to 1.02]
  Follicle Stimulating Hormone | 1.07 [0.78 to 1.46]
  Free Testosterone | 1.71 [1.01 to 2.90]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 7
  Sex Hormone Binding Globulin | 0.25 [0.15 to 0.43]
  Dihydroepiandrosterone Sulfate: number analyzed (Participants) | 9
  Dihydroepiandrosterone Sulfate | 0.87 [0.68 to 1.12]

45. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 9 Day 1
Description: Geometric mean of ratio (Cycle 9 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 9 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 6
Ratio
  Testosterone | 0.38 [0.26 to 0.57]
  Estradiol | 0.56 [0.49 to 0.65]
  Prolactin | 1.19 [0.65 to 2.18]
  LH Serum | 0.72 [0.56 to 0.93]
  Follicle Stimulating Hormone | 0.83 [0.67 to 1.03]
  Free Testosterone | 1.23 [1.08 to 1.40]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 4
  Sex Hormone Binding Globulin | 0.19 [0.09 to 0.39]
  Dihydroepiandrosterone Sulfate | 0.72 [0.51 to 1.00]

46. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 12 Day 1
Description: Geometric mean of ratio (Cycle 12 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 12 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 6
Ratio
  Testosterone | 0.38 [0.14 to 1.04]
  Estradiol: number analyzed (Participants) | 5
  Estradiol | 0.66 [0.32 to 1.37]
  Prolactin | 1.06 [0.72 to 1.57]
  LH Serum | 0.88 [0.59 to 1.32]
  Follicle Stimulating Hormone | 1.02 [0.63 to 1.65]
  Free Testosterone | 1.39 [0.68 to 2.86]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 5
  Sex Hormone Binding Globulin | 0.23 [0.11 to 0.46]
  Dihydroepiandrosterone Sulfate: number analyzed (Participants) | 5
  Dihydroepiandrosterone Sulfate | 0.75 [0.42 to 1.34]

47. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 15 Day 1
Description: Geometric mean of ratio (Cycle 15 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 15 Day 1
Population: Hypogonadism test evaluable population: Male participants who had completed screening, had received at least 1 dose of crizotinib on Cycle 1 Day 1, had at least 1 post baseline visit data for at least total testosterone, free testosterone, SHBG and included male participants of MET amplification and enriched other Cohort following approval of protocol amendment number 21. "N" =participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 4
Ratio
  Testosterone | 0.49 [0.21 to 1.14]
  Estradiol | 1.03 [0.47 to 2.25]
  Prolactin | 1.32 [0.86 to 2.03]
  LH Serum | 0.90 [0.56 to 1.45]
  Follicle Stimulating Hormone | 0.81 [0.53 to 1.22]
  Free Testosterone | 1.71 [0.57 to 5.13]
  Sex Hormone Binding Globulin | 0.24 [0.12 to 0.49]
  Dihydroepiandrosterone Sulfate | 0.76 [0.57 to 0.99]

48. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 18 Day 1
Description: Geometric mean of ratio (Cycle 18 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 18 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 3
Ratio
  Testosterone | 0.32 [0.22 to 0.48]
  Estradiol: number analyzed (Participants) | 2
  Estradiol | 0.55 [0.03 to 8.69]
  Prolactin | 1.64 [1.12 to 2.39]
  LH Serum | 0.69 [0.58 to 0.82]
  Follicle Stimulating Hormone | 0.89 [0.53 to 1.47]
  Free Testosterone | 1.10 [0.42 to 2.91]
  Sex Hormone Binding Globulin: number analyzed (Participants) | 2
  Sex Hormone Binding Globulin | 0.18 [0.07 to 0.45]
  Dihydroepiandrosterone Sulfate | 0.69 [0.20 to 2.35]

49. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 21 Day 1
Description: Geometric mean of ratio (Cycle 21 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 21 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 2
Ratio
  Testosterone | 0.23 [0.09 to 0.60]
  Estradiol: number analyzed (Participants) | 1
  Estradiol | 0.48
  Prolactin | 1.46 [0.62 to 3.41]
  LH Serum | 0.53 [0.12 to 2.42]
  Follicle Stimulating Hormone | 0.77 [0.44 to 1.33]
  Free Testosterone | 1.23 [0.00 to 797.68]
  Sex Hormone Binding Globulin | 0.15 [0.00 to 20.43]
  Dihydroepiandrosterone Sulfate | 0.72 [0.09 to 5.76]

50. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 24 Day 1
Description: Geometric mean of ratio (Cycle 24 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 24 Day 1
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 2
Ratio
  Testosterone | 0.39 [0.00 to 70772.27]
  Estradiol | 0.70 [0.00 to 11581.59]
  Prolactin | 1.13 [0.10 to 12.55]
  LH Serum | 0.69 [0.09 to 5.23]
  Follicle Stimulating Hormone | 0.53 [0.07 to 3.81]
  Free Testosterone: number analyzed (Participants) | 1
  Free Testosterone | 2.35
  Sex Hormone Binding Globulin | 0.20 [0.00 to 33217.86]
  Dihydroepiandrosterone Sulfate | 0.90 [0.48 to 1.66]

51. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 27 Day 1
Description: Geometric mean of ratio (Cycle 27 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 27 Day 1
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 2
Ratio
  Testosterone | 0.46 [0.00 to 61000.31]
  Estradiol | 0.97 [0.00 to 9022.66]
  Prolactin | 1.48 [0.11 to 20.69]
  LH Serum | 0.70 [0.11 to 4.50]
  Follicle Stimulating Hormone | 0.66 [0.06 to 7.53]
  Free Testosterone | 1.86 [0.02 to 147.95]
  Sex Hormone Binding Globulin | 0.24 [0.00 to 22059.61]
  Dihydroepiandrosterone Sulfate | 0.95 [0.24 to 3.78]

52. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at Cycle 30 Day 1
Description: Geometric mean of ratio (Cycle 30 Day 1/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, Cycle 30 Day 1
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 1
Ratio
  Testosterone | 0.16
  Estradiol | 0.38
  Prolactin | 1.14
  LH Serum | 0.85
  Follicle Stimulating Hormone | 0.80
  Free Testosterone | 1.25
  Sex Hormone Binding Globulin | 0.09
  Dihydroepiandrosterone Sulfate | 0.71

53. Primary Outcome: Geometric Mean of Ratio of Total Testosterone, Free Testosterone, Sex Hormone Binding Globulin (SHBG), Luteinizing Hormone, Follicle Stimulating Hormone, Dihydroepiandrosterone Sulfate, Estradiol and Prolactin Levels in Males at End of Treatment
Description: Geometric mean of ratio (End of treatment/Baseline) of hypogonadism parameters (total testosterone, free testosterone, sex hormone binding globulin, luteinizing hormone, follicle stimulating hormone, dihydroepiandrosterone sulfate, estradiol and prolactin) levels in males was analyzed. Data for this outcome measure was planned to be collected for combined RP2D Cohort only, excluding arms of low and high dose escalation cohorts. 95% CI should be interpreted with cautions due to the limited sample size at this time point.
Time Frame: Baseline, End of Treatment (28 days post last dose)
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RP2D Cohort: Crizotinib 250 mg
Number analyzed (Participants) | 5
Ratio
  Testosterone | 0.40 [0.08 to 2.08]
  Estradiol | 0.66 [0.39 to 1.13]
  Prolactin | 1.48 [0.49 to 4.50]
  LH Serum | 0.52 [0.14 to 1.98]
  Follicle Stimulating Hormone | 0.85 [0.26 to 2.72]
  Free Testosterone | 0.62 [0.20 to 1.93]
  Sex Hormone Binding Globulin | 0.64 [0.24 to 1.71]
  Dihydroepiandrosterone Sulfate: number analyzed (Participants) | 4
  Dihydroepiandrosterone Sulfate | 0.41 [0.21 to 0.78]

ADVERSE EVENTS:
Time Frame: Up to maximum of 189 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Groups:
- Itraconazole Interaction Sub-study: Crizotinib 250 mg: Participants received Crizotinib 250 mg (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) capsule/tablet QD from Cycle 1Day1 to Cycle 2 Day1 thereafter 250 mg BID from Cycle 2 Day 2 up to 58 cycles (each cycle 28 days). Participants also received Itraconazole 200 mg QD from Cycle 1 Day 1 to Cycle 1 Day 16.
- Midazolam Interaction Cohort: Crizotinib 250: Participants received Crizotinib 250 mg tablet/capsule (2 capsules/tablet of 100 mg each + 1 capsule/tablet of 50 mg) orally BID from Day 1Cycle 1 up to p to 133 cycles (each cycle 28 days). Participants also received single 2 mg oral dose of Midazolam on Day -7 and another single 2-mg oral dose of Midazolam concurrently with Crizotinib on Cycle 2 Day 1.
Arm/Group | Low Dose Escalation Cohort: Crizotinib 50 mg QD | Low Dose Escalation Cohort: Crizotinib 100 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg QD | Low Dose Escalation Cohort: Crizotinib 200 mg BID | Low Dose Escalation Cohort: Crizotinib 250 mg BID | Low Dose Escalation Cohort: Crizotinib 300 mg BID | High Dose Escalation Cohort: Crizotinib 300 mg QD | High Dose Escalation Cohort: Crizotinib 400 mg QD | High Dose Escalation Cohort: Crizotinib 500 mg QD | High Dose Escalation Cohort: Crizotinib 650 mg QD | High Dose Escalation Cohort: Crizotinib 800 mg QD | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg | RP2D Cohort: Enriched Other: Crizotinib 250 mg | Itraconazole Interaction Sub-study: Crizotinib 250 mg | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin | Midazolam Interaction Cohort: Crizotinib 250
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/8 | 0/7 | 0/8 | 0/6 | 1/6 | 0/5 | 1/3 | 1/6 | 1/9 | 10/53 | 15/85 | 8/41 | 13/48 | 9/18 | 25/154 | 15/66 | 0/18 | 1/18 | 4/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 1/8 | 2/7 | 4/8 | 2/6 | 2/6 | 2/5 | 1/3 | 2/6 | 4/9 | 24/53 | 54/85 | 25/41 | 22/48 | 9/18 | 75/154 | 29/66 | 7/18 | 6/18 | 6/12
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 8/8 | 7/7 | 8/8 | 6/6 | 6/6 | 4/5 | 3/3 | 6/6 | 9/9 | 53/53 | 85/85 | 41/41 | 46/48 | 18/18 | 154/154 | 66/66 | 18/18 | 18/18 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Escalation Cohort: Crizotinib 50 mg QD (N=3) | Low Dose Escalation Cohort: Crizotinib 100 mg QD (N=4) | Low Dose Escalation Cohort: Crizotinib 200 mg QD (N=8) | Low Dose Escalation Cohort: Crizotinib 200 mg BID (N=7) | Low Dose Escalation Cohort: Crizotinib 250 mg BID (N=8) | Low Dose Escalation Cohort: Crizotinib 300 mg BID (N=6) | High Dose Escalation Cohort: Crizotinib 300 mg QD (N=6) | High Dose Escalation Cohort: Crizotinib 400 mg QD (N=5) | High Dose Escalation Cohort: Crizotinib 500 mg QD (N=3) | High Dose Escalation Cohort: Crizotinib 650 mg QD (N=6) | High Dose Escalation Cohort: Crizotinib 800 mg QD (N=9) | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg (N=53) | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg (N=85) | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg (N=41) | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg (N=48) | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg (N=18) | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg (N=154) | RP2D Cohort: Enriched Other: Crizotinib 250 mg (N=66) | Itraconazole Interaction Sub-study: Crizotinib 250 mg (N=18) | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin (N=18) | Midazolam Interaction Cohort: Crizotinib 250 (N=12)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 10 | 8 | 6 | 8 | 1 | 19 | 12 | 0 | 0 | 4
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 11 | 3 | 2 | 0 | 15 | 3 | 0 | 0 | 1
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 2 | 4 | 0 | 7 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 1 | 1 | 10 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic arthritis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 (0)
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fat necrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Low Dose Escalation Cohort: Crizotinib 50 mg QD (N=3) | Low Dose Escalation Cohort: Crizotinib 100 mg QD (N=4) | Low Dose Escalation Cohort: Crizotinib 200 mg QD (N=8) | Low Dose Escalation Cohort: Crizotinib 200 mg BID (N=7) | Low Dose Escalation Cohort: Crizotinib 250 mg BID (N=8) | Low Dose Escalation Cohort: Crizotinib 300 mg BID (N=6) | High Dose Escalation Cohort: Crizotinib 300 mg QD (N=6) | High Dose Escalation Cohort: Crizotinib 400 mg QD (N=5) | High Dose Escalation Cohort: Crizotinib 500 mg QD (N=3) | High Dose Escalation Cohort: Crizotinib 650 mg QD (N=6) | High Dose Escalation Cohort: Crizotinib 800 mg QD (N=9) | RP2D Cohort: ROS1-Positive NSCLC: Crizotinib 250 mg (N=53) | RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg (N=85) | RP2D Cohort: MET Amplification NSCLC: Crizotinib 250 mg (N=41) | RP2D Cohort: ALK-Negative Cohort 1, NSCLC: Crizotinib 250 mg (N=48) | RP2D Cohort: ALK-Negative Cohort 2, NSCLC: Crizotinib 250 mg (N=18) | RP2D Cohort: ALK-Positive Cohort, NSCLC: Crizotinib 250 mg (N=154) | RP2D Cohort: Enriched Other: Crizotinib 250 mg (N=66) | Itraconazole Interaction Sub-study: Crizotinib 250 mg (N=18) | RP2D Cohort: Rifampin Interaction: Crizotinib 250 mg +Rifampin (N=18) | Midazolam Interaction Cohort: Crizotinib 250 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 8 | 14 | 8 | 2 | 2 | 17 | 15 | 4 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 3 | 1 | 14 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 9 | 2 | 2 | 5 | 2 | 26 | 5 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 1 | 6 | 3 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 13 | 2 | 2 | 1 | 13 | 2 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 11 | 4 | 5 | 0 | 9 | 3 | 0 | 0 | 0/0
Syncope (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 2 | 0 | 9 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0/0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 8 | 5 | 3 | 0 | 8 | 3 | 1 | 2 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4 | 3 | 43 | 11 | 6 | 26 | 9 | 92 | 22 | 3 | 10 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 1 | 0 | 12 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 7 | 0 | 1 | 1 | 10 | 3 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 8 | 11 | 7 | 2 | 2 | 8 | 7 | 2 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 3 | 4 | 1 | 19 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3 | 2 | 3 | 3 | 2 | 4 | 4 | 24 | 45 | 10 | 21 | 11 | 68 | 15 | 11 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 25 | 50 | 17 | 17 | 5 | 93 | 32 | 7 | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 6 | 5 | 2 | 3 | 1 | 19 | 4 | 4 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 10 | 5 | 1 | 0 | 12 | 1 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 7 | 1 | 3 | 0 | 17 | 5 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 6 | 3 | 3 | 3 | 2 | 1 | 3 | 3 | 5 | 33 | 49 | 14 | 20 | 10 | 97 | 41 | 10 | 12 | 7
Vomiting (Gastrointestinal disorders) | 2 | 2 | 5 | 4 | 4 | 1 | 3 | 2 | 1 | 2 | 5 | 28 | 35 | 15 | 26 | 9 | 81 | 34 | 8 | 10 | 8
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 3 | 3 | 1 | 14 | 4 | 0 | 0 | 6
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 5 | 4 | 3 | 0 | 16 | 5 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 12 | 1 | 1 | 0 | 7 | 5 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 6 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 3 | 4 | 3 | 3 | 1 | 2 | 2 | 3 | 20 | 35 | 11 | 23 | 8 | 59 | 26 | 8 | 6 | 5
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 2 | 1 | 0 | 14 | 3 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 27 | 49 | 14 | 15 | 4 | 69 | 18 | 3 | 5 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 3 | 6 | 1 | 12 | 5 | 2 | 2 | 0
Pyrexia (General disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 15 | 12 | 2 | 6 | 2 | 34 | 3 | 3 | 3 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 3 | 1 | 7 | 0 | 26 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 5 | 3 | 2 | 12 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 1 | 0 | 7 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 1 | 5 | 4 | 39 | 1 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 11 | 5 | 1 | 1 | 13 | 5 | 1 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 6 | 14 | 5 | 3 | 1 | 19 | 6 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 17 | 19 | 9 | 4 | 0 | 35 | 11 | 3 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 16 | 15 | 10 | 8 | 2 | 30 | 10 | 3 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 11 | 6 | 4 | 1 | 5 | 9 | 3 | 3 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 1 | 1 | 1 | 12 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 5 | 11 | 9 | 2 | 2 | 28 | 5 | 1 | 2 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 6 | 5 | 2 | 1 | 33 | 2 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 4 | 2 | 2 | 4 | 1 | 1 | 2 | 1 | 3 | 16 | 24 | 7 | 9 | 3 | 50 | 20 | 5 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 5 | 3 | 6 | 6 | 2 | 13 | 6 | 4 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 8 | 3 | 1 | 7 | 1 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 9 | 12 | 3 | 2 | 8 | 10 | 3 | 3 | 0 — MedDRA v24.1 was used for RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg group.
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 5 | 2 | 2 | 8 | 4 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 11 | 12 | 3 | 1 | 10 | 11 | 2 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 6 | 5 | 2 | 29 | 10 | 0 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 16 | 4 | 4 | 4 | 22 | 7 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 14 | 12 | 4 | 5 | 32 | 9 | 1 | 2 | 1 — MedDRA v24.1 was used for RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg group.
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 3 | 6 | 3 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 5 | 0 | 20 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 6 | 1 | 6 | 1 | 27 | 3 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 8 | 16 | 7 | 5 | 0 | 12 | 4 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 6 | 1 | 1 | 1 | 8 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 5 | 0 | 15 | 4 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 12 | 2 | 1 | 2 | 11 | 3 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7 | 11 | 2 | 2 | 1 | 18 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 21 | 25 | 9 | 12 | 3 | 65 | 15 | 5 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 19 | 4 | 2 | 0 | 7 | 4 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 15 | 16 | 3 | 7 | 2 | 34 | 8 | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 3 | 2 | 13 | 2 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 1 | 6 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 0 | 13 | 4 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 2 | 6 | 0 | 21 | 3 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 7 | 3 | 2 | 0 | 0 | 18 | 4 | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 1 | 15 | 4 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 3 | 0 | 12 | 3 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 7 | 11 | 6 | 2 | 0 | 26 | 7 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 9 | 1 | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 24 | 7 | 7 | 4 | 24 | 3 | 5 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9 | 2 | 1 | 0 | 10 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 12 | 27 | 10 | 11 | 4 | 34 | 14 | 8 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 1 | 3 | 1 | 10 | 1 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 8 | 3 | 1 | 1 | 4 | 0 | 2 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 6 | 0 | 11 | 2 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 11 | 4 | 2 | 3 | 8 | 1 | 2 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 9 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 1 | 2 | 2 | 5 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 2 | 3 | 1 | 2 | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 5 | 0 | 2 | 1 | 12 | 2 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 5 | 1 | 2 | 0 | 19 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 9 | 4 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 2 | 0 | 17 | 3 | 4 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 15 | 6 | 2 | 2 | 2 | 41 | 5 | 3 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 6 | 4 | 2 | 9 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 19 | 7 | 2 | 0 | 15 | 5 | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 3 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 11 | 7 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 0 | 5 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 6 | 3 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 3 | 3 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 10 | 1 | 2 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 8 | 1 | 1 | 1 | 13 | 2 | 2 | 2 | 1
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal drusen (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual brightness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vitreous degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 19 | 3 | 0 | 0 | 4 | 4 | 3 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 3 | 5 | 2 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 2 | 0 | 4 | 0 | 3 | 2 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral blood blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breakthrough pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 0 | 13 | 2 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0 | 1 | 0 | 8 | 0 | 2 | 0 | 0 — MedDRA v24.1 was used for RP2D Cohort: MET Exon 14 Alterations NSCLC: Crizotinib 250 mg group.
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 9 | 0 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 17 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 5 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 2 | 0 | 4 | 0 | 2 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 5 | 1 | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 4 | 1 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Optic nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site rash (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 7 | 4 | 4 | 3 | 13 | 4 | 2 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 0 | 2 | 4 | 1 | 2 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4 | 1 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Iron binding capacity total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 0 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 4 | 1 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transferrin saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vital dye staining cornea present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 4 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 5 | 0 | 1 | 4 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 4 | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 0 | 8 | 4 | 1 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 6 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 1 | 10 | 3 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 8 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 0 | 7 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 8 | 3 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Visual perseveration (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 5 | 1 | 1 | 8 | 1 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 10 | 4 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 12 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 0 | 0 | 0 | 10 | 2 | 3 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 5 | 3 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 9 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 2 | 2 | 0 | 7 | 1 | 0 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT00585195/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT00585195/SAP_001.pdf